CLINICAL TRIAL: NCT03325387
Title: A Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3305677 in Healthy Subjects
Brief Title: A Study of Multiple Doses of LY3305677 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16619; I8P-MC-OXAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3305677 (Experimental): Escalating doses of LY3305677 administered by subcutaneous (SC) injection
  Interventions: Drug: LY3305677
- Placebo (Placebo Comparator): Saline solution administered by SC injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3305677 — Administered SC
  Arms: LY3305677
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purposes of this study are to determine:

* The safety of LY3305677 and any side effects that might be associated with it.
* How much LY3305677 gets into the bloodstream and how long it takes the body to remove it in healthy participants, including those of Japanese origin.
* The effect LY3305677 has on the body, particularly the effect on blood glucose levels.

This study will last approximately 17 weeks not including screening. Screening is required within 4 weeks prior to start of the study.

This study is for research purposes only and is not intended to treat any medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Women not of child-bearing potential due to surgical sterilization confirmed by medical history or menopause
* Are first-generation Japanese or non-Japanese. First-generation Japanese is defined as the participant, the participant's biological parents, and all of the participant's grandparents are of exclusive Japanese descent and have been born in Japan
* Have a body weight of more than 54 kilograms (kg)

Exclusion Criteria:

* Currently enrolled in a clinical study or have participated in a study within the past 3 months
* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening
* Have history of pancreatitis
* Have known or ongoing psychiatric disorders
* Have undergone bariatric surgery or have used any drugs for weight loss
* Have a history of alcoholism
* Currently smoke more than 10 cigarettes a day

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through 115 days
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3305677 | Days 1 and 29: Predose through 168 hours post dose
  PK: Cmax of LY3305677
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3305677 | Days 1 and 29: Predose through 168 hours post dose
  PK: AUC of LY3305677

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leeds, West Yorkshire, United Kingdom